CLINICAL TRIAL: NCT03652051
Title: A Multicenter, Vehicle-controlled, Randomized Study to Evaluate the Safety, Tolerability, Systemic Pharmacokinetics, and Pharmacodynamics of AZR-MD-001 in Patients With Meibomian Gland Dysfunction (MGD) and Evaporative Dry Eye Disease (DED)
Brief Title: A Multicenter Study Evaluating AZR-MD-001 in Patients With Meibomian Gland Dysfunction and Evaporative Dry Eye Disease (DED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Azura Ophthalmics (Industry)
Collaborators: Syneos Health (Other); Cliantha Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AZ201801
Record Dates: First submitted 2018-08-27; First posted 2018-08-29 (Actual); Results first posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Meibomian Gland Dysfunction; Dry Eye
MeSH Terms: conditions — Meibomian Gland Dysfunction; Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- AZR-MD-001 Low Dose (Experimental): AZR-MD-001 Low Dose will be dosed up to once daily.
  Interventions: Drug: AZR-MD-001 Low Dose
- AZR-MD-001 Mid Dose (Experimental): AZR-MD-001 Mid Dose will be dosed up to once daily.
  Interventions: Drug: AZR-MD-001 Mid Dose
- AZR-MD-001 High Dose (Experimental): AZR-MD-001 High Dose will be dosed up to once daily.
  Interventions: Drug: AZR-MD-001 High Dose
- AZR-MD-001 Vehicle (Sham Comparator): AZR-MD-001 Vehicle will be dosed up to once daily.
  Interventions: Drug: AZR-MD-001 Vehicle

INTERVENTIONS:
Drug: AZR-MD-001 Low Dose — AZR-MD-001 is an ophthalmic ointment
  Arms: AZR-MD-001 Low Dose
Drug: AZR-MD-001 Mid Dose — AZR-MD-001 is an ophthalmic ointment
  Arms: AZR-MD-001 Mid Dose
Drug: AZR-MD-001 High Dose — AZR-MD-001 is an ophthalmic ointment
  Arms: AZR-MD-001 High Dose
Drug: AZR-MD-001 Vehicle — AZR-MD-001 is a vehicle ophthalmic ointment
  Arms: AZR-MD-001 Vehicle

SUMMARY:
AZ201801 is a multicenter study of AZR-MD-001 ointment and AZR-MD-001 vehicle in patients with Meibomian Gland Dysfunction (MGD) and evaporative Dry Eye Disease (DED)

DETAILED DESCRIPTION:
AZ201801 is a multicenter, double-masked, vehicle-controlled, randomized, parallel group study carried out in 2 sequentially overlapping cohorts evaluating the safety, efficacy and tolerability of AZR-MD-001 ointment and AZR-MD-001 vehicle in patients with Meibomian Gland Dysfunction (MGD) and evaporative Dry Eye Disease (DED)

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or older
* Best-corrected visual acuity (BCVA) of 20/40 or better (Snellen equivalent), using the logarithm of the minimum angle of resolution (LogMAR) in each eye
* Evidence of meibomian gland obstruction
* Reported dry eye signs and symptoms within the past 3 months

Exclusion Criteria:

* Uncontrolled ocular disease (except for MGD and dry eye disease/keratoconjunctivitis sicca) or uncontrolled systemic disease
* Glaucoma, ocular hypertension, or intraocular pressure (IOP) in either eye at screening ≥24 mm Hg or has planned insertion/removal of glaucoma filtration shunts/devices during the study
* Corneal abnormality or disorder that impacts normal spreading of the tear film or corneal integrity
* BCVA worse than 20/40 in either eye
* Current use of punctal plugs, anticipated insertion during the study, or a history of punctal cautery in either eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2022-09-14 (Actual); Study Completion 2022-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie L Watson, Principal Investigator — Save Sight Institute
Locations (30):
- Australia (12):
  - Vision Eye Institute, Chatswood, New South Wales
  - Eye Associates, Sydney, New South Wales
  - Sydney Eye Hospital, Sydney, New South Wales
  - School of Optometry and Vision Science, University of New South Wales, Sydney, New South Wales
  - Queensland University of Technology, Brisbane, Queensland
  - Queensland Eye Institute, South Brisbane, Queensland
  - Ophthalmic Trials Australia, Teneriffe, Queensland
  - Eye Laser Specialists, Armadale, Victoria
  - Bendigo Eye Clinic, Bendigo, Victoria
  - Waverley Eye Clinic, Glen Waverley, Victoria
  - Downie Laboratory, Department of Optometry and Vision Sciences, Melbourne, Victoria
  - Deakin University, Waurn Ponds, Victoria
- Canada (16):
  - Seema Eye Care, Calgary, Alberta
  - FYI Doctors, Campbell River, British Columbia
  - VCH Research Institute., Vancouver, British Columbia
  - Ophthalmology, Vancouver, British Columbia
  - Ocean Optometry, Halifax, Nova Scotia
  - Miller Optometry, Halifax, Nova Scotia
  - Prism Eye Institute, Brampton, Ontario
  - Cliantha Research, Mississauga, Ontario
  - Precision Cornea Centre, Ottawa, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - FYI Doctors, Toronto, Ontario
  - Healthpoint, Toronto, Ontario
  - Eyes on Sheppard Clinic, Toronto, Ontario
  - Toronto Eye Care, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - School of Optometry & Vision Science, University of Waterloo, Waterloo, Ontario
- New Zealand (2):
  - University of Auckland, Auckland
  - AucklandEye, Auckland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Watson SL, Jones LW, Stapleton F, Hinds M, Ng A, Tan J, Alster Y, Bosworth C, Rafaeli O, DePuy V; CELESTIAL STUDY Group. Efficacy and safety of AZR-MD-001 selenium sulfide ophthalmic ointment in adults with meibomian gland dysfunction: A vehicle-controlled, randomized clinical trial. Ocul Surf. 2023 Jul;29:537-546. doi: 10.1016/j.jtos.2023.07.002. Epub 2023 Jul 20. PMID 37478969

RESULTS

PARTICIPANT FLOW:
Groups:
- AZR-MD-001 Low Dose: AZR-MD-001 Low Dose was dosed twice weekly.
  AZR-MD-001 Low Dose: AZR-MD-001 is an ophthalmic ointment
- AZR-MD-001 Mid Dose: AZR-MD-001 Mid Dose was dosed twice weekly.
  AZR-MD-001 Mid Dose: AZR-MD-001 is an ophthalmic ointment
- AZR-MD-001 High Dose: AZR-MD-001 High Dose was dosed twice weekly.
  AZR-MD-001 High Dose: AZR-MD-001 is an ophthalmic ointment
- AZR-MD-001 Vehicle: AZR-MD-001 Vehicle was dosed twice weekly.
  AZR-MD-001 Vehicle: AZR-MD-001 is a vehicle ophthalmic ointment
Period: Stage 1
Arm/Group | AZR-MD-001 Low Dose | AZR-MD-001 Mid Dose | AZR-MD-001 High Dose | AZR-MD-001 Vehicle
Started | 9 | 27 | 24 | 16
Completed | 9 | 22 | 16 | 15
Not Completed | 0 | 5 | 8 | 1
Not completed — Adverse Event | 0 | 5 | 7 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Period: Stage 2
Arm/Group | AZR-MD-001 Low Dose | AZR-MD-001 Mid Dose | AZR-MD-001 High Dose | AZR-MD-001 Vehicle
Started (Stage 2 was conducted without including any subjects from Stage 1 to enable Stage 2 to qualify as a confirmatory efficacy study based upon feedback from the FDA at a pre-IND meeting.) | 0 | 82 | 83 | 80
Completed | 0 | 66 | 67 | 74
Not Completed | 0 | 16 | 16 | 6
Not completed — Adverse Event | 0 | 2 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 6 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 11 | 9 | 3

BASELINE CHARACTERISTICS:
Groups:
- Stage 1: AZR-MD-001 Low Dose: AZR-MD-001 Low Dose was dosed twice weekly.
  AZR-MD-001 Low Dose: AZR-MD-001 is an ophthalmic ointment
- Stage 1: AZR-MD-001 Mid Dose; Stage 2: AZR-MD-001 Mid Dose: AZR-MD-001 Mid Dose was dosed twice weekly.
  AZR-MD-001 Mid Dose: AZR-MD-001 is an ophthalmic ointment
- Stage 1: AZR-MD-001 High Dose; Stage 2: AZR-MD-001 High Dose: AZR-MD-001 High Dose was dosed twice weekly.
  AZR-MD-001 High Dose: AZR-MD-001 is an ophthalmic ointment
- Stage 1: AZR-MD-001 Vehicle; Stage 2: AZR-MD-001 Vehicle: AZR-MD-001 Vehicle was dosed twice weekly.
  AZR-MD-001 Vehicle: AZR-MD-001 is a vehicle ophthalmic ointment
- Total: Total of all reporting groups
Arm/Group | Stage 1: AZR-MD-001 Low Dose | Stage 1: AZR-MD-001 Mid Dose | Stage 1: AZR-MD-001 High Dose | Stage 1: AZR-MD-001 Vehicle | Stage 2: AZR-MD-001 Mid Dose | Stage 2: AZR-MD-001 High Dose | Stage 2: AZR-MD-001 Vehicle | Total
Number analyzed (Participants) | 9 | 27 | 24 | 16 | 82 | 83 | 80 | 321
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (18.79) | 42.1 (17.71) | 45.6 (22.02) | 43.6 (20.34) | 52.1 (16.9) | 55.6 (17.2) | 51.9 (18.5) | 53.2 (17.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 11 | 11 | 5 | 51 | 56 | 56 | 196
  Male | 3 | 16 | 13 | 11 | 31 | 27 | 24 | 125
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 5 | 3 | 2 | 10
  Not Hispanic or Latino | 9 | 25 | 22 | 14 | 77 | 80 | 78 | 305
  Unknown or Not Reported | 0 | 2 | 2 | 2 | 0 | 0 | 0 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 10 | 8 | 8 | 16 | 10 | 21 | 77
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0 | 3 | 3 | 1 | 7
  White | 5 | 15 | 14 | 6 | 57 | 64 | 56 | 217
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2 | 2 | 6 | 5 | 2 | 19
Meibomian Glands Yielding Liquid Secretion (Primary Sign Endpoint) [Mean (Standard Deviation); unit: Gland Count (0 to 15)] — Count of the number of open glands on the inferior lid ranging from 0 (no open glands) to 15 (total number of evaluated glands)
  Gland Count (0 to 15) | 2.5 (0.58) | 2.8 (1.26) | 2.9 (1.49) | 2.8 (1.64) | 1.7 (1.4) | 1.9 (1.4) | 1.8 (1.3) | 1.8 (1.3)
OSDI Total Score (Primary Symptom Endpoint) [Mean (Standard Deviation); unit: Total Score (0 to 100)] — The total score on the OSDI ranges from 0 (normal) to 100 (severe disease)
  Total Score (0 to 100) | 25 (7.42) | 23.1 (6.10) | 21.34 (4.86) | 22.64 (7.57) | 25.2 (7.5) | 24.2 (6) | 25 (6.7) | 24.8 (6.7)

OUTCOME MEASURES:

1. Primary Outcome: Meibomian Glands Yielding Liquid Secretion (MGYLS)
Description: Change from Baseline in MGYLS. The MGYLS can range from 0 (abnormal) to 15 (normal)
Time Frame: Value at month 3 minus value at baseline
Measure: Mean (Standard Deviation); unit: Number of Open Glands
Arm/Group | Stage 1: AZR-MD-001 Low Dose | Stage 1: AZR-MD-001 Mid Dose | Stage 1: AZR-MD-001 High Dose | Stage 1: AZR-MD-001 Vehicle | Stage 2: AZR-MD-001 Mid Dose | Stage 2: AZR-MD-001 High Dose | Stage 2: AZR-MD-001 Vehicle
Number analyzed (Participants) | 9 | 27 | 24 | 16 | 82 | 83 | 80
Number of Open Glands | -0.7 (1.56) | 3.41 (0.8) | 3.07 (0.81) | 1.88 (1.38) | 4.2 (0.36) | 3.2 (0.4) | 2.4 (0.34)

2. Primary Outcome: Ocular Surface Disease Index (OSDI) Total Score
Description: Change from Baseline in OSDI Total Score. The OSDI Total Score can range from 100 (highly abnormal) to 0 (Normal)
Time Frame: Value at month 3 minus value at baseline
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Stage 1: AZR-MD-001 Low Dose | Stage 1: AZR-MD-001 Mid Dose | Stage 1: AZR-MD-001 High Dose | Stage 1: AZR-MD-001 Vehicle | Stage 2: AZR-MD-001 Mid Dose | Stage 2: AZR-MD-001 High Dose | Stage 2: AZR-MD-001 Vehicle
Number analyzed (Participants) | 9 | 27 | 24 | 16 | 82 | 83 | 80
Scores on a Scale | 12.93 (4.62) | -8.73 (2.37) | -4.74 (2.41) | -2.34 (4.09) | -7.29 (1.3) | -6.1 (1.3) | -3.8 (1.2)

ADVERSE EVENTS:
Time Frame: 3 months
Description: AEs were classified into system organ class (SOC) and preferred term (PT) using MedDRA version 23.0 or higher. Treatment-emergent adverse events (TEAEs) were defined as events beginning or worsening on or after the planned first dose of study medication.
Arm/Group | Stage 1: AZR-MD-001 Low Dose | Stage 1: AZR-MD-001 Mid Dose | Stage 1: AZR-MD-001 High Dose | Stage 1: AZR-MD-001 Vehicle | Stage 2: AZR-MD-001 Mid Dose | Stage 2: AZR-MD-001 High Dose | Stage 2: AZR-MD-001 Vehicle
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/27 | 0/24 | 0/16 | 0/82 | 0/83 | 0/80
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/27 | 2/24 | 0/16 | 1/82 | 1/83 | 2/80
Other Adverse Events (participants affected / at risk) | 2/9 | 13/27 | 14/24 | 4/16 | 54/82 | 60/83 | 8/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 1: AZR-MD-001 Low Dose (N=9) | Stage 1: AZR-MD-001 Mid Dose (N=27) | Stage 1: AZR-MD-001 High Dose (N=24) | Stage 1: AZR-MD-001 Vehicle (N=16) | Stage 2: AZR-MD-001 Mid Dose (N=82) | Stage 2: AZR-MD-001 High Dose (N=83) | Stage 2: AZR-MD-001 Vehicle (N=80)
pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 (1) | 0 (0) | 0 (0) — pneumonia
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 (0) | 0 (0) | 1 (80) — Pericarditis
Thyroid mass (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 (0) | 0 (0) | 1 (80) — Thyroid mass
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 (0) | 1 (83) | 0 (0) — Post procedural haemorrhage
n intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
ocular toxicity (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 1: AZR-MD-001 Low Dose (N=9) | Stage 1: AZR-MD-001 Mid Dose (N=27) | Stage 1: AZR-MD-001 High Dose (N=24) | Stage 1: AZR-MD-001 Vehicle (N=16) | Stage 2: AZR-MD-001 Mid Dose (N=82) | Stage 2: AZR-MD-001 High Dose (N=83) | Stage 2: AZR-MD-001 Vehicle (N=80)
Application site pain (Eye disorders) | 1 (9) | 12 (32) | 9 (24) | 1 (11) | 14 (16) | 13 (15) | 0 (0) — Application site pain
Lacrimation increased (Eye disorders) | 0 (0) | 4 (32) | 3 (24) | 0 (0) | 9 (9) | 1 (1) | 0 (0) — Lacrimation increased
Punctate keratitis (Eye disorders) | 0 (0) | 1 (32) | 0 (0) | 0 (0) | 8 (8) | 7 (15) | 1 (2) — Punctate keratitis
Vital dye staining cornea present (Eye disorders) | 0 (0) | 1 (32) | 2 (24) | 0 (0) | 5 (7) | 7 (11) | 1 (2) — Vital dye staining cornea present
Eye pain (Eye disorders) | 0 (0) | 3 (32) | 4 (24) | 0 (0) | 5 (5) | 6 (10) | 1 (1) — Eye pain
Eye irritation (Eye disorders) | 0 (0) | 7 (32) | 2 (24) | 0 (0) | 4 (5) | 5 (7) | 2 (3) — Eye irritation
Application site reaction (Eye disorders) | 0 (0) | 1 (32) | 1 (24) | 0 (0) | 4 (5) | 4 (5) | 0 (0) — Application site reaction
Foreign body sensation (Eye disorders) | 1 (9) | 2 (32) | 2 (24) | 2 (11) | 4 (4) | 2 (2) | 1 (1) — Foreign body sensation
Administration site reaction (Eye disorders) | 1 (9) | 2 (32) | 7 (24) | 2 (11) | 4 (4) | 1 (2) | 0 (0) — Administration site reaction
Photophobia (Eye disorders) | 0 (0) | 5 (32) | 3 (24) | 0 (0) | 4 (4) | 1 (1) | 1 (1) — Photophobia
Eye inflammation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 8 (9) | 1 (1) — Eye inflammation
Application site irritation (Eye disorders) | 0 (0) | 2 (32) | 0 (0) | 0 (0) | 2 (2) | 5 (5) | 0 (0) — Application site irritation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-03-19): https://cdn.clinicaltrials.gov/large-docs/51/NCT03652051/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-22): https://cdn.clinicaltrials.gov/large-docs/51/NCT03652051/SAP_001.pdf